CLINICAL TRIAL: NCT00882713
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once- Monthly Administration of Subcutaneous CERA for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anemia
Brief Title: A Study of Once Monthly Subcutaneous Mircera in Dialysis Patients With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21797
Record Dates: First submitted 2009-02-17; First posted 2009-04-16 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- C.E.R.A. (Experimental): Eligible participants will be administered continuous erythropoietin receptor activator (C.E.R.A.[Mircera]) intravenously (IV) every 4 weeks for 44 weeks. The starting dose of 120, 200, or 360 micrograms (mcg) will be based on the dose of epoetin alfa or beta administered in the week preceding the switch to C.E.R.A. Subsequent doses will be adjusted to maintain the individual participant's hemoglobin (Hb) within a range of +/- 1.0 grams per deciliter (g/dL) of the reference hemoglobin (Hb) concentration and between 10.50 and 12.50 g/dL.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Subcutaneous injection every 4 weeks (starting dose of 120, 200 or 360 micrograms, based on previous ESA therapy)
  Other Names: C.E.R.A.

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of once monthly administration of subcutaneous Mircera for the maintenance of hemoglobin levels in dialysis patients with chronic renal anemia. Patients will receive subcutaneous Mircera at a starting dose of 120, 200 or 360 micrograms every 4 weeks, calculated from the last weekly dose of epoetin or darbepoetin alfa previously administered. Subsequent doses will be adjusted to maintain hemoglobin levels within the target range. Treatment duration is 56 weeks, and the target sample size is 200 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* regular long-term hemodialysis or peritoneal dialysis, with same mode of dialysis for >=3 months;
* continuous iv maintenance epoetin alfa therapy with same dosing interval during previous 2 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension;
* significant acute or chronic bleeding;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Morocco (9):
  - Agadir
  - Casablanca
  - FÉS
  - Khouribga
  - Marrakesh
  - Méknés
  - Rabat
  - Salé
  - Tangier

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 participants were enrolled in this study conducted from 12 February 2009 to 25 October 2010 at 28 study sites in Morocco.
Pre-assignment Details: Of 202 participants, 8 participants did not complete the stability verification period (SVP) of 4 weeks. Overall, 194 participants entered dose titration period (DTP) of 16 weeks.
Groups:
- C.E.R.A.: Eligible participants were administered continuous erythropoietin receptor activator (C.E.R.A.) intravenously (IV) every 4 weeks for 44 weeks. The starting dose of C.E.R.A. (120, 200, or 360 micrograms [mcg]) was based on the dose of epoetin alfa or beta administered in the week preceding the switch to C.E.R.A. Subsequent doses were adjusted to maintain the individual participant's hemoglobin (Hb) value within a range of +/- 1.0 grams per deciliter (g/dL) of the reference Hb concentration and between 10.50 and 12.50 g/dL.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 194
Completed | 172
Not Completed | 22
Not completed — Adverse Event | 2
Not completed — Death | 3
Not completed — Administrative reasons | 4
Not completed — refused treatment/withdrew consent | 4
Not completed — Blood transfusion | 2
Not completed — Insufficient therapeutic response | 3
Not completed — Failure to return | 2
Not completed — Other - Reasons | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who have been treated with at least one dose of the study drug and a safety follow-up, whether withdrawn prematurely or not.
Groups:
- C.E.R.A.: Eligible participants were administered C.E.R.A. intravenously (IV) every 4 weeks for 44 weeks. The starting dose of C.E.R.A. (120, 200, or 360 micrograms [mcg]) was based on the dose of epoetin alfa or beta administered in the week preceding the switch to C.E.R.A. Subsequent doses were adjusted to maintain the individual participant's hemoglobin (Hb) value within a range of +/- 1.0 grams per deciliter (g/dL) of the reference Hb concentration and between 10.50 and 12.50 g/dL.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
Age, Continuous [Median (Full Range); unit: years] | 51.5 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 118

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Mean Hemoglobin Concentration Within +/- 1 g/dL of Their Reference Hb and Between 10.5 and 12.5 g/dL During Efficacy Evaluation Period
Description: The percentage of participants who maintained their mean Hb concentration within +/- 1 g/dL of their reference Hb and between 10.5 and 12.5 g/dL during the Efficacy Evaluation Period (EEP) is reported. The EEP was from Week 17 to Week 24. The reference Hb was calculated from the mean of Hb concentrations based upon the Hb assessments at Weeks -4, -3, -2, -1, and 0.
Time Frame: EEP (Week 17 to Week 24)
Population: The per-protocol (PP) population included all participants from the intention-to-treat (ITT) population, who fulfilled inclusion/exclusion criteria as per the study protocol. A total of 123 participants were included in the PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 123
Percentage of participants | 52.0 [42.8 to 61.1]

2. Secondary Outcome: Mean Change in Hemoglobin Concentration Between Reference (Stability Verification Period) and the Efficacy Evaluation Period
Description: Mean change in Hb concentration between reference SVP and the EEP is reported. The SVP was at Weeks -3, -2, -1, and EEP was from Week 17 to Week 24. Participants received epoetin alfa or beta during SVP.
Time Frame: SVP (Weeks -3, -2, -1) and EEP (Week 17 to Week 24)
Population: ITT population included all the participants who had received at least one dose of C.E.R.A. (Week 0) and for whom data for at least one follow-up variable (laboratory data, adverse events, etc.) was available. Out of 194 participants, one was excluded from the ITT population due to missing Hb measurement and C.E.R.A drug after Week 0.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- C.E.R.A.: Eligible participants were administered C.E.R.A. intravenously (IV) every 4 weeks for 44 weeks. The starting dose of C.E.R.A. (120, 200, or 360 mcg) was based on the dose of epoetin alfa or beta administered in the week preceding the switch to C.E.R.A. Subsequent doses were adjusted to maintain the individual participant's hemoglobin (Hb) value within a range of +/- 1.0 g/dL of the reference Hb concentration and between 10.50 and 12.50 g/dL.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 193
g/dL | 0.48 (1.05)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within the Range of 10.5-12.5 g/dL Throughout the EEP
Description: Percentage of participants maintaining Hb concentration within the range of 10.5-12.5 g/dL throughout the EEP is reported. The EEP was from Week 17 to Week 24.
Time Frame: EEP (Week 17 to Week 24)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 193
Percentage of participants | 60.6 [53.4 to 67.6]

4. Secondary Outcome: Mean Time Spent By Participants With Hemoglobin Range of 10.5-12.5 g/dL During the EEP
Description: Mean time spent by participants in Hb range of 10.5-12.5 g/dL during the EEP is reported. The EEP was from Week 17 to Week 24.
Time Frame: EEP (Week 17 to Week 24)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 193
Days | 35.1 (19.85)

5. Secondary Outcome: Number of Participants With Any Adverse Events or Serious Adverse Events
Description: An adverse event (AE) is untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAEs) is with any of the following outcomes: Death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, and congenital anomaly.
Time Frame: Up to Week 52
Population: Safety population included all participants who have been treated with at least one dose of the study drug and completed a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: Participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
Participants
  Any AEs | 39
  Any SAEs | 19

6. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustment During DTP and EEP
Description: Percentage of participants requiring any dose adjustment during DTP (Week 1 to Week 16) and EEP (Week 17 to Week 24) is reported. The dose adjustments (increase or decrease) were required: if a single Hb concentration was either > or = 13 g/dL or < or = 9 g/dL; if the difference of 2 consecutive Hb concentrations was > or =2 g/dL; if the values of scheduled Hb assessments on the day of administration of C.E.R.A. and on the previous study visit were both out of range of 10.5 to 11.5 g/dL, the difference between the reference value (mean of Hb concentrations based on the Hb assessments at Weeks -4, -3, -2, -1, and 0) and the most recent value was >1 g/dL; if the values of the scheduled Hb assessments on the day of administration of C.E.R.A. and on the previous study visit were both out of the range 10 to 12 g/dL. Dose adjustment could be made at any time at the discretion of the clinician if clinically warranted.
Time Frame: DTP (Week 1 to Week 16) and EEP (Week 17 to Week 24)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 193
Percentage of participants
  Dose adjustment during DTP (n = 193) | 56
  Dose adjustment during EEP (n = 185) | 34.6

7. Secondary Outcome: Incidences of Red Blood Cell Transfusions During the C.E.R.A. Treatment Phase
Description: Red Blood Cells (RBCs) transfusions were given during the treatment period in case of medical need. Blood transfusions occurred during the DTP, EEP, and during the long term safety period (LTSP) were reported.
Time Frame: Up to Week 52
Population: as for outcome 5
Measure: Number; unit: Number of RBCs transfusion
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
Number of RBCs transfusion
  During DTP | 3
  During EEP | 1
  During LTSP | 2

8. Secondary Outcome: Mean Hemoglobin Levels Over Time
Description: The Hb levels were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: Safety population included all participants who have been treated with at least one dose of the study drug and completed a safety follow-up, whether withdrawn prematurely or not. Number of participants with available data at specified period is denoted by 'n'.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
g/dL
  Hb at Week 0 (n = 194) | 11.2 (0.58)
  Hb at Week 8 (n = 184) | 11.7 (1.35)
  Hb at Week 16 (n = 175) | 11.8 (1.21)
  Hb at Week 24 (n = 180) | 11.8 (1.14)
  Hb at Week 32 (n = 177) | 11.8 (1.23)
  Hb at Week 40 (n = 162) | 11.8 (1.23)
  Hb at Week 48 (n = 168) | 11.6 (1.20)

9. Secondary Outcome: Mean Hematocrit Levels Over Time
Description: The hematocrit (HCT) levels were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
Proportion of red blood cells in blood
  HCT at Week 0 (n = 194) | 0.34 (0.02)
  HCT at Week 8 (n = 184) | 0.36 (0.04)
  HCT at Week 16 (n = 175) | 0.36 (0.04)
  HCT at Week 24 (n = 180) | 0.36 (0.04)
  HCT at Week 32 (n = 177) | 0.36 (0.04)
  HCT at Week 40 (n = 163) | 0.36 (0.04)
  HCT at Week 48 (n = 170) | 0.35 (0.04)

10. Secondary Outcome: Mean Albumin Levels Over Time
Description: The albumin levels were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: Safety population included all participants who have been treated with at least one dose of the study drug and a safety follow-up, whether withdrawn prematurely or not. Out of 194, one participant was excluded from the ITT population due to missing hemoglobin measurement and C.E.R.A medication after Week 0.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 193
g/L
  Albumin at Week 0 (n = 193) | 43.1 (8.61)
  Albumin at Week 8 (n = 139) | 41.0 (6.65)
  Albumin at Week 16 (n = 130) | 41.3 (6.44)
  Albumin at Week 24 (n = 128) | 40.2 (6.19)
  Albumin at Week 32 (n = 116) | 39.9 (6.12)
  Albumin at Week 40 (n = 108) | 40.4 (6.47)
  Albumin at Week 48 (n = 147) | 39.9 (7.26)

11. Secondary Outcome: Mean White Blood Cells and Thrombocytes Over Time
Description: The white blood cells (WBCs) and thrombocyte levels were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
10^9 cells/L
  WBCs at Week 0 (n = 194) | 6.5 (1.75)
  WBCs at Week 8 (n = 153) | 6.5 (2.00)
  WBCs at Week 16 (n = 137) | 6.3 (1.71)
  WBCs at Week 24 (n = 138) | 6.4 (2.00)
  WBCs at Week 32 (n = 129) | 6.3 (1.81)
  WBCs at Week 40 (n = 123) | 6.3 (1.78)
  WBCs at Week 48 (n = 153) | 6.5 (1.74)
  Thrombocytes at Week 0 (n = 194) | 213.9 (68.51)
  Thrombocytes at Week 8 (n = 153) | 207.5 (65.64)
  Thrombocytes at Week 16 (n = 137) | 202.5 (58.62)
  Thrombocytes at Week 24 (n = 138) | 200.5 (55.74)
  Thrombocytes at Week 32 (n = 129) | 208.6 (69.50)
  Thrombocytes at Week 40 (n = 123) | 206.1 (68.12)
  Thrombocytes at Week 48 (n = 153) | 204.7 (68.95)

12. Secondary Outcome: Mean Phosphate and Potassium Levels Over Time
Description: The phosphate and potassium levels were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milimole/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
milimole/L
  Phosphate at Week 0 (n = 194) | 1.7 (0.57)
  Phosphate at Week 8 (n = 139) | 1.7 (0.76)
  Phosphate at Week 16 (n = 131) | 1.7 (0.75)
  Phosphate at Week 24 (n = 130) | 1.7 (0.70)
  Phosphate at Week 32 (n = 116) | 1.6 (0.56)
  Phosphate at Week 40 (n = 110) | 1.4 (0.44)
  Phosphate at Week 48 (n = 148) | 1.6 (0.61)
  Potassium at Week 0 (n = 194) | 5.3 (0.91)
  Potassium at Week 8 (n = 139) | 5.4 (0.95)
  Potassium at Week 16 (n = 131) | 5.4 (0.99)
  Potassium at Week 24 (n = 130) | 5.5 (1.02)
  Potassium at Week 32 (n = 117) | 5.5 (0.92)
  Potassium at Week 40 (n = 110) | 5.5 (0.93)
  Potassium at Week 48 (n = 146) | 5.3 (0.92)

13. Secondary Outcome: Mean Creatinine, Iron, and Total Iron Binding Capacity Levels Over Time
Description: The mean creatinine, iron, and total iron binding capacity (TIBC) levels over time were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromole/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
micromole/L
  Creatinine at Week 0 (n = 194) | 775.7 (477.80)
  Creatinine at Week 8 (n = 139) | 692.5 (502.86)
  Creatinine at Week 16 (n = 130) | 676.1 (490.80)
  Creatinine at Week 24 (n = 130) | 683.7 (472.92)
  Creatinine at Week 32 (n = 117) | 670.2 (477.22)
  Creatinine at Week 40 (n = 110) | 674.8 (488.26)
  Creatinine at Week 48 (n = 149) | 699.6 (444.93)
  Iron at Week 0 (n = 194) | 15.9 (8.04)
  Iron at Week 8 (n = 139) | 15.1 (7.49)
  Iron at Week 16 (n = 129) | 15.1 (6.74)
  Iron at Week 24 (n = 130) | 14.3 (5.08)
  Iron at Week 32 (n = 116) | 14.9 (5.50)
  Iron at Week 40 (n = 110) | 15.6 (5.59)
  Iron at Week 48 (n = 148) | 15.2 (5.92)
  TIBC at Week 0 (n = 194) | 44.5 (11.46)
  TIBC at Week 8 (n = 137) | 44.2 (10.90)
  TIBC at Week 16 (n = 126) | 44.8 (12.40)
  TIBC at Week 24 (n = 123) | 43.7 (11.10)
  TIBC at Week 32 (n = 116) | 44.1 (11.33)
  TIBC at Week 40 (n = 110) | 42.6 (10.58)
  TIBC at Week 48 (n = 147) | 44.0 (10.37)

14. Secondary Outcome: Mean C-Reactive Protein Levels Over Time
Description: The mean C-Reactive Protein (CRP) Levels over time were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: miligrams/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
miligrams/L
  CRP at Week 0 (n = 190) | 6.9 (8.84)
  CRP at Week 8 (n = 139) | 7.9 (8.98)
  CRP at Week 16 (n = 130) | 8.6 (11.19)
  CRP at Week 24 (n = 127) | 9.3 (13.87)
  CRP at Week 32 (n = 112) | 7.1 (7.33)
  CRP at Week 40 (n = 109) | 7.2 (7.77)
  CRP at Week 48 (n = 140) | 7.4 (8.76)

15. Secondary Outcome: Mean Ferritin Levels Over Time
Description: The mean ferritin levels over time were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
mcg/L
  Ferritin at Week 0 (n = 194) | 547.6 (896.63)
  Ferritin at Week 8 (n = 138) | 522.2 (772.16)
  Ferritin at Week 16 (n = 129) | 517.6 (639.09)
  Ferritin at Week 24 (n = 128) | 508.6 (577.75)
  Ferritin at Week 32 (n = 116) | 522.6 (874.94)
  Ferritin at Week 40 (n = 110) | 562.8 (984.72)
  Ferritin at Week 48 (n = 148) | 505.6 (770.48)

16. Secondary Outcome: Mean Transferrin Saturation Levels Over Time
Description: The mean transferrin saturation (TSAT) levels over time were recorded for each participant at enrolment and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of Transferrin Saturation
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 194
Percentage of Transferrin Saturation
  TSAT at Week 0 (n = 194) | 37.3 (20.16)
  TSAT at Week 8 (n = 136) | 35.0 (16.38)
  TSAT at Week 16 (n = 125) | 36.0 (18.45)
  TSAT at Week 24 (n = 123) | 34.9 (18.24)
  TSAT at Week 32 (n = 115) | 35.4 (14.72)
  TSAT at Week 40 (n = 110) | 38.0 (15.66)
  TSAT at Week 48 (n = 147) | 36.5 (17.56)

17. Secondary Outcome: Mean Change From Baseline in Pulse Rate Over Time
Description: Mean change in pulse rate was defined as the difference between mean pulse rate at Baseline and following visits (Weeks 8, 16, 24, 32, 40, and 48).
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: Safety population included all participants who have been treated with at least one dose of the study drug and completed a safety follow-up, whether withdrawn prematurely or not. Participants with available data at the time of evaluation were analyzed. Number of participants with available data at specified period is denoted by 'n'.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 190
beats per minute
  Week 8 (n = 175) | 0.37 (6.21)
  Week 16 (n = 175) | 0.02 (6.61)
  Week 24 (n = 173) | 0.30 (6.86)
  Week 32 (n = 173) | 0.40 (6.97)
  Week 40 (n = 174) | 0.52 (8.24)
  Week 48 (n = 190) | 0.76 (8.69)

18. Secondary Outcome: Mean Change From Baseline in Blood Pressure Over Time
Description: Mean change in blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) before and after dialysis was defined as the difference between mean blood pressure at Baseline and following visits (Weeks 8, 16, 24, 32, 40, and 48).
Time Frame: Baseline (Week 0) and Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 191
millimeter of mercury
  SBP before dialysis at Week 8 (n = 189) | 1.15 (14.41)
  SBP before dialysis at Week 16 (n = 185) | -0.78 (13.08)
  SBP before dialysis at Week 24 (n = 182) | -0.58 (13.14)
  SBP before dialysis at Week 32 (n = 181) | -1.28 (14.68)
  SBP before dialysis at Week 40 (n = 175) | 0.27 (13.24)
  SBP before dialysis at Week 48 (n = 191) | -0.52 (13.72)
  SBP after dialysis at Week 8 (n = 185) | 1.68 (12.62)
  SBP after dialysis at Week 16 (n = 181) | 0.48 (12.94)
  SBP after dialysis at Week 24 (n = 178) | 0.60 (13.10)
  SBP after dialysis at Week 32 (n = 177) | 0.40 (14.45)
  SBP after dialysis at Week 40 (n = 171) | 1.22 (11.97)
  SBP after dialysis at Week 48 (n = 187) | 1.63 (13.97)
  DBP before dialysis at Week 8 (n = 189) | -0.77 (11.85)
  DBP before dialysis at Week 16 (n = 185) | -1.87 (11.00)
  DBP before dialysis at Week 24 (n = 182) | -1.58 (11.56)
  DBP before dialysis at Week 32 (n = 181) | -2.08 (9.56)
  DBP before dialysis at Week 40 (n = 175) | -1.35 (10.23)
  DBP before dialysis at Week 48 (n = 191) | -0.90 (10.72)
  DBP after dialysis at Week 8 (n = 185) | -0.40 (9.04)
  DBP after dialysis at Week 16 (n = 181) | -0.11 (10.35)
  DBP after dialysis at Week 24 (n = 178) | -0.90 (9.47)
  DBP after dialysis at Week 32 (n = 177) | -1.07 (8.56)
  DBP after dialysis at Week 40 (n = 171) | -1.50 (8.95)
  DBP after dialysis at Week 48 (n = 187) | -1.21 (10.11)

19. Secondary Outcome: Mean Change From Baseline in Weight Over Time
Description: Mean change in weight was defined as the difference between mean weight at Baseline and following visits (Week 16 and Week 48).
Time Frame: Week 16 and Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 191
kilogram
  Week 16 (n = 185) | -0.20 (3.17)
  Week 48 (n = 191) | 0.06 (3.21)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Safety population included all participants who have been treated with at least one dose of the study drug and completed a safety follow-up, whether withdrawn prematurely or not.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 19/194
Other Adverse Events (participants affected / at risk) | 15/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=194)
Angina pectoris (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1 — General disorders and administration site conditions
Drug effect decreased (General disorders) | 1 — General disorders and administration site conditions
Arteriovenous fistula site infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3
Fluid overload (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=194)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Bronchitis (Infections and infestations) | 11
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.